CLINICAL TRIAL: NCT00919477
Title: Protocol for the Specified Clinical Experience Investigation on the Single Use of Casodex® Tablet 80 mg
Acronym: CAMON
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OJP-CAS-2009/1; CAS002
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Casodex; Monotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To gather information on the safety of monotherapy of Casodex® tablets 80 mg, targeting prostate cancer patients who have no history of having received treatment by either endocrine therapy (including surgical castration).

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients who have no history of receiving endocrine therapy (including surgical castration), and who plan to undergo Casodex® tablets monotherapy for not less than 12 months

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prostate cancer patients who have no history of having received treatment by either endocrine therapy (including surgical castration)
Sampling Method: Probability Sample
Enrollment: 712 (Actual)
Dates: Start 2009-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Adverse event incidence | Time since starting Casodex monotherapy, monthly

SECONDARY OUTCOMES:
improvement of prostate cancer using Tumor marker PSA | Time since starting Casodex monotherapy, monthly
Maintenance of sexual function | At 3 months since starting Casodex monotherapy,

CONTACTS AND LOCATIONS:
Locations (160):
- Japan (160):
  - Research Site, Houmei, Aichi-ken
  - Research Site, Inuyama, Aichi-ken
  - Research Site, Kasugai, Aichi-ken
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Okazaki, Aichi-ken
  - Research Site, Toyohashi, Aichi-ken
  - Research Site, Toyota, Aichi-ken
  - Research Site, Akita, Akita
  - Research Site, Ōdate, Akita
  - Research Site, Hirosaki, Aomori
  - Research Site, Asahi, Chiba
  - Research Site, Funahashi, Chiba
  - Research Site, Ichihara, Chiba
  - Research Site, Ichikawa, Chiba
  - Research Site, Narashino, Chiba
  - Research Site, Sakura, Chiba
  - Research Site, Imabari, Ehime
  - Research Site, Matsuyama, Ehime
  - Research Site, Niihama, Ehime
  - Research Site, Uwajima, Ehime
  - Research Site, Chikushino-shi, Fukuoka
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Iizuka, Fukuoka
  - Research Site, Kasuga, Fukuoka
  - Research Site, Kitakyushu, Fukuoka
  - Research Site, Kurume, Fukuoka
  - Research Site, Yukuhashi, Fukuoka
  - Research Site, Aizu-Wakamatsu, Fukushima
  - Research Site, Fukushima, Fukushima
  - Research Site, Gifu, Gifu
  - Research Site, Ibi, Gifu
  - Research Site, Kani, Gifu
  - Research Site, Minokamo, Gifu
  - Research Site, Mizunami, Gifu
  - Research Site, Ōgaki, Gifu
  - Research Site, Sekimachi, Gifu
  - Research Site, Yamagata, Gifu
  - Research Site, Yourou, Gifu
  - Research Site, Isesaki, Gunma
  - Research Site, Kiryū, Gunma
  - Research Site, Numata, Gunma
  - Research Site, Ohta, Gunma
  - Research Site, Takasaki, Gunma
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Eniwa, Hokkaido
  - Research Site, Kushiro, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Sunagawa, Hokkaido
  - Research Site, Tomakomai, Hokkaido
  - Research Site, Akashi, Hyōgo
  - Research Site, Katou, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Takarazuka, Hyōgo
  - Research Site, Hitachi, Ibaraki
  - Research Site, Mito, Ibaraki
  - Research Site, Sashima, Ibaraki
  - Research Site, Toride, Ibaraki
  - Research Site, Tsuchiura, Ibaraki
  - Research Site, Hakusan, Ishihawa
  - Research Site, Hizume, Iwate
  - Research Site, Ichinoseki, Iwate
  - Research Site, Kamaishi, Iwate
  - Research Site, Miyako, Iwate
  - Research Site, Morioka, Iwate
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Zentrsuji, Kagawa-ken
  - Research Site, Minamisatsuma, Kagoshima-ken
  - Research Site, Atsugi, Kanagawa
  - Research Site, Chigasaki, Kanagawa
  - Research Site, Ebina, Kanagawa
  - Research Site, Kawasaki, Kanagawa
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Yamato, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Yokosuka, Kanagawa
  - Research Site, Kochi, Kochi
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Nantan, Kyoto
  - Research Site, Inabe, Mie-ken
  - Research Site, Tsu, Mie-ken
  - Research Site, Matsushima, Miyagi
  - Research Site, Natori-shi, Miyagi
  - Research Site, Sendai, Miyagi
  - Research Site, Shiogama, Miyagi
  - Research Site, Tagajō-shi, Miyagi
  - Research Site, Isahaya, Nagasaki
  - Research Site, Nagasaki, Nagasaki
  - Research Site, Sasebo, Nagasaki
  - Research Site, Ikoma, Nara
  - Research Site, Kashiba, Nara
  - Research Site, Nara, Nara
  - Research Site, Gosen, Niigata
  - Research Site, Tsubame, Niigata
  - Research Site, Nakatsu, Oita Prefecture
  - Research Site, Kurashiki, Okayama-ken
  - Research Site, Okayama, Okayama-ken
  - Research Site, Habikino, Osaka
  - Research Site, Ibaraki, Osaka
  - Research Site, Ikeda, Osaka
  - Research Site, Izumisano, Osaka
  - Research Site, Kaizuka, Osaka
  - Research Site, Kishiwada, Osaka
  - Research Site, Matsubara, Osaka
  - Research Site, Minoo, Osaka
  - Research Site, Motiguchi, Osaka
  - Research Site, Neyagawa, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Ōsaka-sayama, Osaka
  - Research Site, Sakai, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Toyonaka, Osaka
  - Research Site, Yao, Osaka
  - Research Site, Asagiri, Saitama
  - Research Site, Hidaka, Saitama
  - Research Site, Kawagoe, Saitama
  - Research Site, Koshigaya, Saitama
  - Research Site, Kumagaya, Saitama
  - Research Site, Saitama, Saitama
  - Research Site, Sayama, Saitama
  - Research Site, Hamada, Shimane
  - Research Site, Fuji, Shizuoka
  - Research Site, Fujieda, Shizuoka
  - Research Site, Hamamatsu, Shizuoka
  - Research Site, Izu, Shizuoka
  - Research Site, Shimizu, Shizuoka
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Ashikaga, Tochigi
  - Research Site, Tokushima, Tokushima
  - Research Site, Yoshinogawa, Tokushima
  - Research Site, Adachi City, Tokyo
  - Research Site, Arakawa City, Tokyo
  - Research Site, Chiyoda City, Tokyo
  - Research Site, Edogawa City, Tokyo
  - Research Site, Katsushika-ku, Tokyo
  - Research Site, Koutou, Tokyo
  - Research Site, Minato, Tokyo
  - Research Site, Musashino, Tokyo
  - Research Site, Nakano City, Tokyo
  - Research Site, Nishitōkyō, Tokyo
  - Research Site, Oota, Tokyo
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Setagaya City, Tokyo
  - Research Site, Shibuya City, Tokyo
  - Research Site, Shinagawa, Tokyo
  - Research Site, Shinjyuku, Tokyo
  - Research Site, Sumida City, Tokyo
  - Research Site, tabashi City, Tokyo
  - Research Site, Tachikawa, Tokyo
  - Research Site, Toshima City, Tokyo
  - Research Site, Tottori-shi, Tottori
  - Research Site, Kurobe-shi, Toyama
  - Research Site, Takaoka, Toyama
  - Research Site, Toyama, Toyama
  - Research Site, Wakayama, Wakayama
  - Research Site, Yachi, Yamagata
  - Research Site, Yamagata, Yamagata
  - Research Site, Kai, Yamanashi
  - Research Site, Nirasaki, Yamanashi